CLINICAL TRIAL: NCT03900663
Title: Nutritional Status and Body Composition of Children in Relation to Mode of Delivery and Feeding in the First 2 Years of Life
Brief Title: Effect Mode of Delivery and Feeding on Body Composition and Nutritional Status of Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MR Rassmy, Pediatric Resident, Assiut University
Other Study IDs: Delivery,feeding,child obesity
Record Dates: First submitted 2019-03-21; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breast fed infants
  Interventions: Device: Anthropometric measures
- Formula fed infants
  Interventions: Device: Anthropometric measures
- vaginally delivered infants
  Interventions: Device: Anthropometric measures
- Infants delivered by caesarean section
  Interventions: Device: Anthropometric measures

INTERVENTIONS:
Device: Anthropometric measures — Measure body weight , height , chest circumference , mid upper arm circumference,skin fold thickness , head circumference

SUMMARY:
* Feeding and growth during infancy have been associated with later life body mass index.
* Breastfeeding seems to have a small but consistent protective effect against obesity in children.
* The Cholesterol content of human milk is 6-fold greater than that of the standard infant formulas.
* Infants delivered by caesarean section may be at increased risk of childhood obesity and adulthood obesity.

DETAILED DESCRIPTION:
* Previous guidelines recommended that infants who are exclusively breast fed for the first 6 months of life, with particular solid foods gradually introduced from 6 months associated with lower childhood fat mass.
* The stated reason for discouraging introduction of solids to infant before 4 months include the risk of excessive weight gain, vulnerability of the gut to infection and increased susceptibility to the development of allergic disease.
* Infants whose dietary pattern was most similar to feeding guidelines, with high frequencies of fresh fruit and vegetables, home prepared foods and breast milk, gained weight and skin fold thickness more rapidly from 6 to12 months than other infants, independent of milk feeding, age of introduction of solids and maternal factors.
* Exclusively breastfed infants had significantly higher Total Cholesterol (TC) level and Low density Lipoprotein level (LDL) and lower High density lipoprotein level (HDL) as compared to mixed-fed infants in the first 6 months of life.
* Exclusive breast feeding seems to have a protective effect against some risk factors for cardiovascular disease in later life, as those who exclusively breastfed had lower level of plasma low density lipoprotein (LDL) cholesterol conc., higher level of high density lipoprotein (HDL) and lower LDL/HDL ratio than those bottle fed.
* Early weaning is related to rapid weight gain in infancy, and this may have implication for childhood obesity.
* Vaginally delivered children are colonised with bacterial strains from the mothers' vagina during delivery in contrast to children delivered by CS, and these differences seem to persist throughout infancy.
* The gut microbiota may have a role in energy harvesting, hence inoculation with maternal microbiota through vaginal delivery may be protective for childhood overweight compared with delivery by CS.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sexes
* Infants from 2 to 3 years
* Breast fed or formula fed or mixed fed infants

Exclusion Criteria:

* Children less than 2 and more than 3 years ago.
* Children having family history of chronic illness
* Children having family history of metabolic
* Children fed cow milk or buffalo milk.
* Infants delivered preterm.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From out patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Obesity | Through one year
  Body mass index (BMI) kg/m2

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harit D, Faridi MM, Aggarwal A, Sharma SB. Lipid profile of term infants on exclusive breastfeeding and mixed feeding: a comparative study. Eur J Clin Nutr. 2008 Feb;62(2):203-9. doi: 10.1038/sj.ejcn.1602692. Epub 2007 Feb 28. PMID 17327867
- [Background] Goldani HA, Bettiol H, Barbieri MA, Silva AA, Agranonik M, Morais MB, Goldani MZ. Cesarean delivery is associated with an increased risk of obesity in adulthood in a Brazilian birth cohort study. Am J Clin Nutr. 2011 Jun;93(6):1344-7. doi: 10.3945/ajcn.110.010033. Epub 2011 Apr 20. PMID 21508088
- [Background] Ravelli AC, van der Meulen JH, Osmond C, Barker DJ, Bleker OP. Infant feeding and adult glucose tolerance, lipid profile, blood pressure, and obesity. Arch Dis Child. 2000 Mar;82(3):248-52. doi: 10.1136/adc.82.3.248. PMID 10685933